CLINICAL TRIAL: NCT02212249
Title: Soluble VE-cadherin and VE-cadherin Antibody in Sclerodermic Sclerosis
Acronym: Sclerocadh1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2014-A00186-41
Record Dates: First submitted 2014-04-23; First posted 2014-08-08 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Primary Raynaud Disease; Systemic Sclerosis
Keywords: soluble VE-cadherin; antibody; systemic slerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systemic sclerosis (Active Comparator): patients with systemic sclerosis
  Interventions: Biological: soluble Ve cadherin
- primary raynaud disease (Sham Comparator): patients with primary raynaud disease
  Interventions: Biological: soluble Ve cadherin

INTERVENTIONS:
Biological: soluble Ve cadherin — dosage of soluble VE cadherine in each arms

SUMMARY:
Ve-cadherin is expressed in endothelial cells. Systemic slerosis is a rare auto-immune disease with a endothelial dysfunction. This study is to evaluated the level of soluble VE-cadherin and VE-cadherin antibody in patients with systemic slerosis.

ELIGIBILITY:
Inclusion Criteria:

* group 1: systemic sclerosis
* group 2: raynaud primary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Level of soluble Ve-cadherin and antibody VE-cadherin with ELISA TEST in Scleroderma group versus Primary Raynaud's Phenomenon | At 30 days average
  Level of human sVE and antibody VE-cadherin in blood will be determined by ELISA test in both groups Scleroderma and Primary Raynaud's Phenomenon.
  The methodology of dosage of sVE is based on the pattern:WO/2008/062314 The methodolody of the dosage of antibody VE-cadherin is based on the pattern WO/2012/136820 .
  Group Scleroderma (N=60) versus Primary Raynaud's Phenomenon (N=20). Shapiro test.

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France